Identifiers: NCT05380180

Brief Title: Enhancing Quality of Life for Older Adults With and Without Mild Cognitive

Impairment (MCI) Through Social Engagement Over Video Technology

Document Date: Sept 4, 2023

## **Statistical Analysis Plan**

To measure the main effects of the intervention on primary and secondary outcomes, irrespective of the cognitive status, the OneClick intervention Group will be compared to the Waitlist group at (i) mid-assessment (4 weeks) compared with the baseline assessment, and (ii) post-assessment (8 weeks) compared with baseline assessment. In addition, we will perform a separate analysis of covariance with age and cognitive ability (MoCA and Logical Memory - Delayed Recall) as covariates. We plan to implement an intent-to-treat analysis where all participants who were allocated to either the intervention or waitlist group will be included in the analysis, regardless of the number of sessions attended or their completion of assessments.